CLINICAL TRIAL: NCT06450652
Title: Feasibility, Safety, and Effectiveness of Chinese Herbal Medicine for T2DM Patients With Comorbid Metabolic Syndrome: A Single-arm Pilot Study
Brief Title: CHM for T2DM & MetS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Hong Kong Baptist University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/23-24/0397
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes Mellitus With Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chinese Herbal Medicine granules (Experimental)
  Interventions: Drug: Chinese Herbal Medicine granules

INTERVENTIONS:
Drug: Chinese Herbal Medicine granules — The intervention will be a 4 weeks of Chinese Herbal Medicine (CHM) granules, which will consist of six Chinese herbs. Subjects will take one sachet orally, twice daily after meals for 4 weeks. Way of taking CHM granules is as follow: Add 100ml boiling water into a cup, then pour one pack of granules into the cup and soap it for 2-3 mins. Stir until the granules completely dissolve before drinking.

SUMMARY:
This is a single-arm design. A total of 15 Type 2 Diabetes Mellitus (T2DM) patients with comorbid Metabolic Syndrome (MetS) will be recruited from community. The intervention will be a 4-week of Chinese Herbal Medicine granules treatment, which will consist of six Chinese herbs. The primary outcome measure will be fasting plasma glucose and blood pressure. Secondary outcome measures including changes of anthropometric data (body mass index, waist-to-hip ratio), lipid panels (total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein), HbA1C, Framingham Stroke Risk Score (FSRS), Audit of diabetes-dependent quality of Life (ADDQoL), International Physical Activity Questionnaire Short Form (IPAQ-SF), daily step count and physiological parameters from wearable watch, dietary record, retinal and sublingual vein imaging, concurrent medications and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30-75y.
* Diagnosed with Type 2 diabetes no more than 5 years.
* Having current prehypertension (systolic blood pressure 130-139 mmHg or diastolic blood pressure 85-89mmHg), or with a history of hypertension (systolic blood pressure 140-159mmHg or diastolic blood pressure 90-99mmHg).
* Diagnosed with Metabolic Syndrome according to Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition) from Chinese Diabetes Society. People who meet 3 of the following diagnostic criteria or more can be diagnosed as Metabolic Syndrome: (a)Abdominal obesity: waist circumference ≥ 90cm for male and ≥ 85cm for female; (b) Hyperglycemia: Fasting blood glucose ≥ 6.1mmol/L or 2-hour postprandial glucose ≥ 7.8mmol/L and/or those who have been diagnosed with hyperglycemia and in treatment; (c) Hypertension: blood pressure ≥ 130/85mmHg and/or those who have been diagnosed with hypertension and in treatment; (d) Fasting triglyceride ≥ 1.70mmol/L; (e) Fasting HDL-C < 1.04mmol/L.
* Diagnosed with Accumulation of phlegm and dampness pattern or Intertwined phlegm and blood stasis pattern based on Traditional Chinese Medicine (TCM) theory.
* Stable vital signs and with sufficient sensorimotor and language competency for completing assessments.

Exclusion Criteria:

* Allergic history to Chinese herbal drugs or a known allergy to the ingredients of the CHM.
* Diagnosed with type 1 diabetes, steroid-induced diabetes, gestational diabetes, or specific types of diabetes.
* Diabetes accompanied by severe complications such as diabetic nephropathy, diabetic ketoacidosis, etc.
* Secondary obesity (e.g., secondary to pituitary inflammation, tumor, etc.).
* Secondary hypertension (e.g., pheochromocytoma, renal hypertension, etc.).
* Secondary hyperlipidemia (e.g., hypothyroidism, nephrotic syndrome, etc.).
* Experienced at least one day of diarrhea in the past 7 days.
* With previous stroke history.
* With unconsciousness, aphasia, and cognitive dysfunction.
* With severe heart, liver, or kidney disease or bleeding disorders, or with other serious diseases (e.g. cancer, dementia, etc.).
* Pregnancy or lactation female.
* Had joined other clinical trial within past 4 weeks.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose (FPG) | Baseline, week 2, week 4, week 8.
  FPG will be determined by taking a blood sample from participants who have fasted for 8-12 hours.
Blood pressure | Baseline, week 2, week 4, week 8.
  Blood pressure was measured thrice, after a 10 min rest, using a standard digital sphygmomanometer.

SECONDARY OUTCOMES:
Framingham Stroke Risk Score (FSRS) | Baseline, week 2, week 4, week 8.
  The Framingham Stroke Risk Score (FSRS) combines stroke risk factors (sex, age, systolic blood pressure, high-density lipoprotein level, total cholesterol level, smoking, diabetes) to predict 10-year probability of stroke.
Audit of diabetes-dependent quality of Life (ADDQoL) | Baseline, week 4, week 8.
  The ADDQOL consists of two overview items; one measures generic overall QoL and a further 19 items are concerned with the impact of diabetes on specific aspects of life. The 19 life domains are as follows: leisure activities, working life, local or long-distance journeys, holidays, physical health, family life, friendships and social life, close personal relationships, sex life, physical appearance, self-confidence, motivation to achieve things, people's reactions, feelings about the future, financial situation, living conditions, dependence on others, freedom to eat, and freedom to drink. Lower scores reflect poorer QoL. Finally, a mean weighted impact score (ADDQOL score) is calculated for the entire scale across all applicable domains.
International Physical Activity Questionnaire Short Form (IPAQ-SF) | Baseline, week 2, week 4, week 8.
  IPAQ-SF has been recommended as a cost-effective method to assess physical activity. IPAQ-SF records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate- intensity activity such as leisure cycling, 3) walking, and 4) sitting. It requires participants to recall the number of days and time spent on different intensity of activities in last 7 day.
Anthropometric assessment, lipid panels, HbA1C | Baseline, week 2, week 4, week 8.
  Anthropometric indices such as body height (BH), body weight (BW), waist circumference (WC) and hip circumference (HC) were measured. Body mass index [(BMI) = BW (kg)/BH (m)2] and waist-to-hip ratio [(WHR) = WC (cm)/HC (cm)] will be calculated. Lipid panels (total cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein) will be assessed before and after treatment period. Hemoglobin A1c test, as known as HbA1c, measure the amount of blood glucose attached to hemoglobin, indicating the average blood glucose level for the last two to three months. For diabetic patients, an ideal HbA1c level is 48mmol/mol (6.5%) or below.
Physiological parameters and dietary records | Baseline, week 2, week 4, week 8.
  Wearable watch will be used to record patients' daily step count and physiological parameters. Patients' diet will be assessed by 3-day weighed dietary records (two non-consecutive weekdays and one weekend day).
Adverse events | Baseline, week 2, week 4, week 8.
  All adverse events (AEs), defined as any adverse events that occur from the beginning of the participant's enrollment to the end of the trial, regardless of whether there is a causal relationship with the received treatments, that occur in the trial will be recorded.